CLINICAL TRIAL: NCT06790290
Title: Phase 2, Randomized, Double-blind, Active-controlled Study Evaluating the Safety and Immunogenicity of IVT PCV-25 in Healthy Infants Administered With the WHO Expanded Programme on Immunization 3+0 Vaccine Schedule
Brief Title: Phase 2 Trial to Evaluate Safety and Immunogenicity of Inventprise's (IVT) 25-valent Pneumococcal Conjugate Vaccine (IVT PCV-25) in Healthy Infants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inventprise Inc. (Industry)
Collaborators: University of the Philippines-National Health Institute_Doña Nena Health Center (Unknown); Health Index Multispecialty Clinic (Unknown); Grand Centennial Homes Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVT 121
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-04

CONDITIONS: Pneumococcal Disease, Invasive
Keywords: Vaccine; Healthy Volunteer
MeSH Terms: conditions — Pneumococcal Infections | interventions — D-Worm

STUDY DESIGN:
Intervention Model Description: Subjects are randomized in four groups, 1:1:1:1, each receiving 3 doses of one of three vaccine formulations or comparator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Low dose) (Experimental): Infant participants will receive three 0.5mL dose of IVT PCV-25 Formulation B administered by intramuscular injection on Day 1, 29 and 57
  Interventions: Biological: Formulation B
- Group B (High dose) (Experimental): Infant participants will receive three 0.5mL dose of IVT PCV-25 Formulation C administered by intramuscular injection on Day 1, 29 and 57
  Interventions: Biological: Formulation C
- Group C (Hybrid dose) (Experimental): Infant participants will receive three 0.5mL dose of IVT PCV-25 Formulation D administered by intramuscular injection on Day 1, 29 and 57
  Interventions: Biological: Formulation D
- Group D (Comparator) (Active Comparator): Infant participants will receive three 0.5mL dose of Prevnar20 administered by intramuscular injection on Day 1, 29 and 57
  Interventions: Biological: Prevnar20

INTERVENTIONS:
Biological: Formulation B — IVT PCV-25
  Arms: Group A (Low dose)
Biological: Formulation C — IVT PCV-25
  Arms: Group B (High dose)
Biological: Formulation D — IVT PCV-25
  Arms: Group C (Hybrid dose)
Biological: Prevnar20 — 20 valent pneumococcal conjugate vaccine
  Arms: Group D (Comparator)

SUMMARY:
Phase 2 trial to evaluate safety and immunogenicity of Inventprise's (IVT) 25-valent pneumococcal conjugate vaccine (IVT PCV-25) in Healthy Infants

DETAILED DESCRIPTION:
A Phase 2 multicenter, randomized, active-controlled, double-blind study to evaluate safety and immunogenicity of a 3-dose intramuscular (IM) regimen of three formulations of IVT PCV-25, a 25 valent conjugated pneumococcal vaccine with adjuvant. Infant participants will be randomized in a 1:1:1:1 ratio to receive 3 IM injections of one IVT PCV-25 formulation or the active comparator (Prevnar 20) at 4-week intervals (at approximately 6, 10 and 14 weeks of age) with routine infant vaccines administered on the same day as IVT PCV-25/Prevnar 20.

ELIGIBILITY:
Inclusion Criteria: Participants who meet all the following criteria may be included in the study:

1. Age 42 to 56 days, inclusive, at the time of Dose 1
2. Good general health status, as determined by medical history, physical examination, vital signs, and clinical judgment
3. Product of normal full-term pregnancy (37 to 42 weeks' gestation)
4. Birth weight ≥ 2000 g
5. Length and weight ≥ -2 standard deviations (SD) for age and sex, according to the Philippine national child growth standards (see Appendix 1)
6. Willingness of parent/guardian for the child to attend all protocol visits and to have all protocol-required procedures
7. Provision of written informed consent by legally acceptable representative

Exclusion Criteria: Participants who meet any of the following criteria will be excluded from the study:

1. Congenital abnormality or serious chronic disorder requiring treatment or likely to affect normal growth or development
2. Any condition that may increase risk of study participation or interfere with interpretation of study results
3. Immunodeficiency or chronic administration (> 14 consecutive days) of immunosuppressant or other immune-modifying drugs (see details in Section 6.6.2), including systemic glucocorticoids, within 6 months before Day 1 (topical, intra- articular, or inhaled glucocorticoids permitted)
4. History of sepsis or pneumonia
5. History of anaphylaxis or angioedema
6. History of severe reaction to immunization
7. Known hypersensitivity to any of the ingredients in either IVT PCV-25 or Prevnar 20
8. Contraindication to any concomitant vaccine or to Prevnar 20, according to each vaccine's product information
9. Prior receipt of a licensed or investigational pneumococcal vaccine
10. Prior receipt of any diphtheria, tetanus, pertussis, Hib, or polio vaccine
11. Prior receipt of > 1 dose of HepB vaccine
12. Receipt of HepB vaccine at age ≥ 30 days
13. Receipt of an inactivated vaccine within 14 days before Day 1 or planned receipt through Day 85 other than as described in Section 6.6.1 and Section 6.6.3
14. Receipt of a live vaccine within 28 days before Day 1 or planned receipt through Day 85 other than as described in Section 6.6.1 and Section 6.6.3
15. Receipt of blood transfusion or blood products before Day 1 or planned receipt through Day 85
16. Receipt of any other IP before Day 1
17. Planned elective hospitalization or surgical procedure through the end of the study
18. Family member of employee of Inventprise, vendors, or research sites associated with the study
19. Any medical, psychiatric, or social condition, or occupational or other responsibility of the parent/guardian that, in the judgment of the Investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or an ability to provide informed consent

Temporary Delay Criteria: administration of IVT PCV-25 / Prevnar20 will be delayed for any participant who meets any of the following criteria:

1. Receipt of any inactivated vaccine within 14 days or any live vaccine within 28 days
2. Febrile illness (eg, temperature ≥ 38.0°C) or other acute illness within 48 hours
3. Any other signs or symptoms or medication use that could inhibit the proper vaccine administration of the IP or interpretation of diary data

Ages: 42 Days to 56 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 421 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with reactogenicity events for 7 days after Doses 1, 2, and 3 | 7 days after Doses 1,2,3
  To assess the safety and tolerability of 3 formulations of IVT PCV-25 administered at 6, Percentage of Participants with Reactogenicity Events 7 days after Doses 1,2,3
Percentage of participants with adverse events (AEs) from Dose 1 to 28 days after Dose 3 | From Dose 1 to 28 days after Dose 3
  To assess the safety and tolerability of 3 formulations of IVT PCV-25 administered at 6, 10, and 14 weeks of age
Percentage of participants with medically attended AEs (MAAEs) from Dose 1 to 6 months after Dose 3 | From Dose 1 to 6 months after Dose 3
  To assess the safety and tolerability of 3 formulations of IVT PCV-25 administered at 6, 10,and 14 weeks of age
Percentage of participants with newly diagnosed chronic medical conditions (NDCMCs) from Dose 1 to 6 months after Dose 3 | From Dose 1 to 6 months after Dose 3
  To assess the safety and tolerability of 3 formulations of IVT PCV-25 administered at 6, 10, and 14 weeks of age
Percentage of participants achieving serotype-specific immunoglobulin G (IgG) concentration of ≥ 0.35 µg/mL at 28 days after each dose | from Dose 1 to 6 months after Dose 3
  To assess the safety and tolerability of 3 formulations of IVT PCV-25 administered at 6, 10, and 14 weeks of age

SECONDARY OUTCOMES:
Percentage of participants achieving serotype-specific immunoglobulin G (IgG) concentration of ≥ 0.35 µg/mL at 28 days after each dose | 28 days after each dose
  To assess the humoral immunogenicity of 3 formulations of IVT PCV-25 administered at 6, 10, and 14 weeks of age
Ratio of geometric mean concentrations (GMCs) of serotype-specific IgG, comparing each IVT PCV-25 formulation to Prevnar 20 at 28 days after each dose | 28 days after each dose
  To assess the humoral immunogenicity of 3 formulations of IVT PCV-25 administered at 6, 10, and 14 weeks of age
Ratio of geometric mean titers (GMTs) of serotype-specific functional antibody measured by opsonophagocytic assay (OPA), comparing each IVT PCV-25 formulation to Prevnar 20 at 28 days after Dose 3 | 28 days after each dose
  To assess the humoral immunogenicity of 3 formulations of IVT PCV-25 administered at 6, 10, and 14 weeks of age

OTHER OUTCOMES:
GMCs of concomitant vaccine antibodies at 28 days after Dose 3 | 28 days after Dose 3
  To assess the humoral immunogenicity of vaccines administered concomitantly with IVT PCV-25
Percentage of participants achieving an antibody concentration threshold | 28 days after Dose 3
  To assess the humoral immunogenicity of vaccines administered concomitantly with IVT PCV-25
Number of days on systemic antibiotic treatment/days on study | Day 1 to 6 months after Dose 3
  To evaluate antibiotic use after administration of IVT PCV-25 administered at 6, 10, and 14 weeks of age
Proportion of participants receiving systemic antibiotic treatment from Day 1 to 6 months after Dose 3 | Day 1 to 6 months after Dose 3 administered
  To evaluate antibiotic use after administration of IVT PCV-25 administered at 6, 10, and 14 weeks of age
Incidence of S pneumoniae serotype determination by polymerase chain reaction (PCR) assay in isolates collected from any participant with a pneumococcal infection during the study | Dose 1 to 6 months after Dose 3
  To determine serotypes of any breakthrough S pneumoniae

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Inventprise Inc.
Locations (3):
- Philippines (3):
  - Health Index Multispecialty Clinic, Bacoor, Cavite
  - Grand Centennial Homes Clinic, Kawit, Cavite
  - University of the Philippines-National Health Institute_Doña Nena Health Center, Pasay, National Capital Region

IPD SHARING:
Plan to Share IPD: No